CLINICAL TRIAL: NCT02501252
Title: Effectiveness and Acceptability of Availing Skilled Birth Attendance (SBA) Services Through Community Reproductive Health Nurses (CORN) to a Household Level at Rural Communities of Ethiopia A Cluster Randomized Controlled Community Trial in Gedeo Zone, SNNPR
Brief Title: Effectiveness and Acceptability of Availing Skilled Birth Attendance (SBA) Services Through Community Reproductive Health Nurses (CORN) to a Household Level at Rural Communities of Ethiopia; A Cluster Community Trial in Gedeo Zone, SNNPR
Acronym: CORN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilla University (Other)
Collaborators: Ethiopian Public Health Institute (Other Government); Ministry of Health, Ethiopia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: RPC674
Record Dates: First submitted 2015-07-14; First posted 2015-07-17 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Maternal Care Patterns
Keywords: Community; Skilled birth attendance; Rural; Ethiopia

STUDY DESIGN:
Intervention Model Description: CORN were assigned into three arms namely: HP, HC and control arms
Oversight: Data Monitoring Committee: No

ARMS (3):
- CORN Based at health post (Experimental): Trained CORN based at health post will provide SBA and other RH services on demand at health post or household levels on an outreach bases.
  Interventions: Procedure: trained midwives and nurses working in the community to provide skilled SBA services
- CORN Based at health center (Active Comparator): Trained CORN based at health center, but working in the community in an outreach basis will provide SBA and other RH services
  Interventions: Procedure: trained midwives and nurses working in the community to provide skilled SBA services
- Control (No Intervention): will be composed of a randomly selected comparable controls clusters. Control clusters (arm) will be similar with the other two arms (groups) except for the intervention.

INTERVENTIONS:
Procedure: trained midwives and nurses working in the community to provide skilled SBA services — After the completion of all the necessary preparations, trained CORNs will be deployed for ten months in their respective study sites (arms) to provide the required RH services at home, community and health posts.
  Arms: CORN Based at health center; CORN Based at health post

SUMMARY:
Rationale: Every year, 287,00 million women, and 3.1 million neonates continue to die, and the majority of these deaths have been identified as being avoidable. A proxy indicator of Millennium Development Goal (MDG) 5, birth with skilled attendance is low in Sub-Saharan Africa(47%) and the lowest (13%) is for Ethiopia, with the greatest number of maternal deaths. The Ethiopia health system has established a vast network of health infrastructure that extends to rural areas with the establishment of over 15,000 health posts and deployment of over 30,000 health extension workers throughout the country. Although these unprecedented situations made health services more accessible than ever, it is yet to be exploited for improving rural women's access to clean and safe delivery and postpartum care. Lack of usage of delivery care in the country is related not only to accessibility but also acceptability of the services. In fact, the vast majority of women with home deliveries saw institutional delivery as "unnecessary" and a "non-customary practice". Therefore, instituting an innovative, culturally sensitive, and practically amenable strategy, deployment of CORNs for example might be the best remedy, in this case.

Objective: To evaluate the effectiveness and acceptability of availing Home based Skilled Birth Attendance (SBA) Services through Community Reproductive Health Nurses (CORN) in rural communities of Ethiopia.

Study design: Cluster Randomized Controlled Community Trial that will be conducted in four phases.

Study population: Study participants will be all pregnant women who will give birth at home and health facility (including health post) during the study period.

Intervention: The study will be conducted in four phases as discussed below. During the first (preparatory) phase, sensitization of relevant stakeholders and recruitment of trainees will be conducted. In the second phase, formative and baseline assessment as well as training of CORNs will take place. In the third phase, which will be actual intervention phase, deployment of CORNs in their respective study site will be done and in the final phase, final evaluation and dissemination of study findings will be done. The intension behind deploying CORNs to the grassroots level is just to give a backup skilled delivery and other MNH services to poor rural mothers who have difficult of accessing modern health facilities for various reasons; it has no any intention to promote or encourage home deliveries or replace institutional deliveries. Perhaps it will help to assimilate rural mothers to modern health facilities Main study parameters/endpoints: The main study end point is percentage of skilled birth attendance which is very low in local and national level. In addition secondary study parameters are percentage changes of maternal & related services uptakes. These include focused Antenatal; care (ANC), long term family planning, Prevention of Mother to Child Transmission of HIV (PMTCT) and postnatal care.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: the burden and risks associated with participation to the study is very minimal. To mention few; physical examinations (Leopold manoeuvre) or the routine investigations of pregnancy this will be anonymous except for the CORNs keeping the principles of shared confidentiality in mind. Similarly all questionnaires or medical charts will be kept confidential. All CORNs will obtain intensive training on ethical principles that will help to minimize any physical and physiological discomfort associated with participation, the risks associated with the investigation treatment.

The study period and Budget: the study will be carried out in a total of 18 months which holds a period from the development of protocol to the terminal evaluation and submission of reports. The overall study budget will be 99, 987.95 USD (Ninety nine thousands, nine hundred eighty seven dollars and ninety five cents

DETAILED DESCRIPTION:
Introduction Every year, 287,000 women die during pregnancy or childbirth, and 6.9 million children die before reaching their fifth birthday. Almost all these deaths occur in developing countries where mothers, children and newborns lack access to basic health care. While child mortality rates have declined in recent decades, 19,000 mothers still mourn the loss of a child each and every day - an unthinkable number of heartbreaks. This is especially tragic since most of these deaths could be prevented at a modest cost.

On the other hand, majority of maternal and newborn deaths are caused by complications or conditions that could be prevented or more effectively managed through inexpensive, low-technology measures. Majority of maternal and new born care deaths were followed by unskilled delivery attended at home. A study conducted in Basra about reasons reported by women who delivered at home for preferring home delivery have shown that social support and privacy was the predominant reason given by 98.2% of the women who had home delivery of their present child. Fear of interventions and repeated examinations at hospitals was the concern of 71.9% of the women who preferred home delivery. About 17.5% had an unplanned home delivery as a result of quick labor or the security situation did not allow transfer to hospital.

On the other hand, recent evidences illustrated that maternal deaths can be reduced with the posting of midwives (skilled attendant) if they have needed skills, supervision, and back-up . Evidences obtained from Bangladesh in 2004 suggested that, programme to create a cadre of skilled birth attendants for home births was launched by the Government . Accordingly, task-shifting seems to have yielded beneficial results and important insights into human resources planning for safe motherhood in the country. Another similar study by Ray AM on the impact of maternal mortality interventions using traditional birth attendants and village midwives showed that village midwives contribute to positive programme outcomes.

The presence of a skilled provider during childbirth and the immediate postpartum/newborn period is the single most critical intervention in saving the lives of women and newborns . The skilled provider can assist in normal deliveries and also manage or stabilize and refer for complications; all of which are critical interventions in reducing maternal and newborn mortality. The proportion of women who delivered with the assistance of a skilled birth attendant is one of the proxy indicators in meeting the fifth MDG. In almost all countries where health professionals attend more than 80% of deliveries, Maternal Mortality Rate (MMR)is below 200 per 100,000 live births [11]. However, birth with skilled attendance was low in Southern Asia (40%) and SSA (47%), the two regions with the greatest number of maternal deaths.

Though the program has addressed majority of the health problems at grass root level, maternal and child morbidity/ mortality rates of the nation is still one of the highest in the world. This is mainly attributable to the competency level of the rural health extension workers to provide cross-cutting maternity services on top of the deep rooted cultural, social and economic problems of the rural community. For example, a recent study in Tigray Region of Ethiopia showed that even if the HEWs have contributed substantially to the improvement in women's utilization of family Planning (FP), ANC and HIV testing, their contribution to the improvement in health facility delivery, postnatal check up and use of iodized salt seems insignificant.

In addition to doubts in the skill of the rural Health Extension Worker (HEW), they are also expected to discharge several additional roles and responsibilities along with maternity related services. Moreover, they are not able and encouraged to attend skilled birth delivery services to mothers, rather they are expected to identify the problem and refer to next higher level health facility which are inaccessible (geographically, socially, economically...etc) to the rural community. This will definitely impend better utilization of modern maternity services.

Current study findings in Ethiopia shows that skilled delivery service utilization is very low. Only 13% of the women who had a live birth in preceding five years of the 2011 survey were assisted by a skilled health worker and 12% were delivered in health facilities although this represented an improvement from 6.2% in 2000. This rate is in the lowest bound by sub-Saharan Africa standard. Skilled assistance at delivery estimated to increase at a low pace of 5.6% per annuum and, with this pace, the proportion that will be attended by skilled workers predicted at 21% by 2015. Multivariate analysis suggests rural women, uneducated, and poor were less likely to deliver in health institutions.(13) The major attributable reasons identified are geared towards the level of knowledge about maternity services, cultural influences and low perceived benefit of service utilization.

According to a study on trends in maternal health in Ethiopia 2012, Women who did not deliver in health facilities were asked the reasons for not doing so. The Ethiopian Demographic and Health Survey (EDHS) 2011 data revealed that the two outstanding reasons were "not necessary" and "not customary", as reported by 61.4% and 29.6%, of them respectively. These were followed by place too far/lack of transportation (14.4%). Other reasons were reported by a tiny portion of the women. Only very few (2.1%) blamed service cost as a reason for not delivering in health facilities. Notably, the reporting of these reasons follow similar pattern both in the urban and rural areas. Strikingly, about two-third of the urban women who did not deliver in health facilities said it was not necessary and 17% said it was not customary.

Mothers' reply of "not necessary" and "not customary implies the fact that they need someone very closer to be with them. According to the findings of couple of studies in North West and South-East Ethiopia, (60.9%) of mothers gave brth at home just needing for closer attention by family members, 57.7% said delivering at home is a usual experience, 33.4% said labor was short/urgent, 21.6% said they did not have any problem to go to health facilities, and 14.0% said influence from family members were the reasons for giving birth at home.

What is more is, even if the number and distribution of health workers, particularly nurses, in the country has made progressive improvement, the country is still far behind to achieving maternal and child health related MDGs as the health service utilization rate is by far below the minimum set by the WHO which is a paradox to the above achievements.

Therefore, what can we learn at this stage is that a novel, culturally sensitive and socially acceptable strategy that can overcome the shortcomings and limitations of the above facts must have to come in place if the nation is to achieve the MDGs and the health related Growth and transformation plan. May availing SBA services to the community (household) level through the deployment of Community Reproductive Health Nurses (CORN) at Kebele (the smallest village level administrative unit of Ethiopian government system) level be helpful to fill the majority of these gaps overlooked yet?

2. RESEARCH QUESTIONS

* How effective is availing Home based SBA services by CORN in increasing births attended by skilled birth Attendants?
* What is the level of acceptability for availing Home based SBA services by the service providers, health service managers and the general community(clients)?
* What are the added advantages of deploying Skilled birth Attendants (CORN) who can provide SBA and other MNH services at household levels in strengthening the health extension program of Ethiopia?
* What are the added advantages of deploying Skilled Birth Attendants (CORN) in improving the SBA and other Reproductive Health (RH) services utilization?

  3. OBJECTIVE General Objective: To evaluate the effectiveness and acceptability of availing Home based Skilled Birth Attendance (SBA) Services through Community Reproductive Health Nurses (CORN) in rural communities of Ethiopia.

Primary Specific Objective

* To determine the effect of availing home based SBA services on utilization
* To examine the programmatic and socio-cultural acceptability of home based delivery of SBA services Secondary Objectives
* To determine the effect of the skilled Birth Attendants(CORN) on other RH services utilization.
* To describe the effect of the Skilled Birth Attendants (CORN) in strengthening the Ethiopian Rural Health Extension Program.

  4. METHODS Study design

This study is a two arm (pre-test, post test) Cluster Randomized Controlled Community Trial that will be conducted in four phases. The two arms are:

Arm one : CORNs based at health center will be trained to provide skilled birth attendance and other RH services on demand at household levels on an outreach bases.

Arm two : CORNs will be based and living in the community at health post /kebele/ level to provide SBA services either at the health post or house hold levels.

Interventions of the first arm will be tested for effectiveness and acceptability against the baseline finding. A baseline evaluation and formative assessment using qualitative methods will also be conducted to document the situation of health service utilization and socio-cultural barriers affecting skilled birth attendances at all of the study sites. This will serve as a pretest data for the intervention and control sites. By applying similar techniques and tools, post test data will be collected at the end of the study at all the three arms. The main variable for comparisons in pretest post test data is the coverage of deliveries attended by SBAs in the two arms, be it by CORNS or using the existing facility based service delivery. Data will be collected from health institutions and the community within the study area. The difference between pretest and post test indicators within and between the intervention arms will be measured to the effect of the intervention in changing the SBA service uptake.

Study Area and period The study will be conducted in three districts of Gedeo Zone ,Southern Region of Ethiopia with population of density of 650 per Sq. Kms.,. The Region is one of the nine Regions in the country which makes 20% of national population. Gedeo Zone is one of the highly populated areas in Ethiopia and in Africa at large. The Zonal town, Dilla, is located some 365 and 92 Kms away from the national and regional capitals, Addis Ababa and Hawassa respectively.

Dilla University is one of the public Universities in Ethiopia situated in the study site. Currently the University has 12 faculties and three Colleges including College of Health Sciences and a Referral Hospital. The maternal health service coverage and utilization of Gedeo zone is one of the lowest in the country (7, 29).

This implementation study is expected to take around one and half year as from the time of securing project grant to terminal evaluation and dissemination.

In the health institutions (health centers and health posts), the health record data on SBA service coverage (institutional delivery, ANC and PNC) will be checked as the secondary source of information. Primary data in relation to the barriers and facilitating factors will be collected using semi-structured questionnaire for service providers. In-depth interviews and focus group discussions will also be conducted, among the service providers, health service managers and the community separately to get insights in to the perceptions, barriers and facilitators of skilled birth attendance services as well as the extent and acceptability of deploying CORN.

Sample size and sampling procedure A cluster randomized community trial proposes to assess the effectiveness of deploying CORNs to advance skilled birth attendance (delivery). A previous Demographic and health Survey (DHS) 2011 study showed that proportion of subjects who had an assisted delivery was 4% in rural settings. According to the health sector development plan IV of the country, it has been planned to increase the proportion of assisted delivery from 18.4% to 62% at the end of 2014/15 fiscal year. Hence, a pro-grammatically similar and important difference of 58% is expected after the deployment of CORNs.

Assuming the Level of significance = 5%, Power = 80%, Type of test = two-sided Based on the above stated assumptions, the initial sample size required per group is 94. To estimate the sample size for a cluster randomized trial, we needed an estimate of the degree of clustering at the practice level, which was available from a previous randomized trial of postnatal care . Using the approach of a previous study, and taking the inter-practice correlation coefficient to be 0.005 as indicated in that trial, we inflated the sample size by 2.45 times from a non-cluster randomized trial considering the potential cluster design effect. This yielded an estimated sample size in each group to be 230. Hence total sample size required for the two arm trial is 460.

A sample size of 460 households, 230 in each arm, is sufficient to detect a clinically important difference of 58% between groups in assisting delivery by deploying CORN using a two-tailed z-test of proportions between two groups with 80% power and a 5% level of significance. This 58% difference represents a 62% assisted delivery by CORNs and 4% assisted delivery without CORN or routine standard of community care. All other secondary outcomes yielded a sample size of much lower than the one stated above. Hence, for the sake of sample adequacy, for the analysis to be carried out for both primary and secondary outcome, the maximum sample size (490) is considered.

Study Participants Study participants will be All pregnant women who will give birth at home and health facility (including health post) during the study period.

Husbands, grandmothers and health workers ( for the qualitative formative assessment)

The Intervention The study will be conducted in four phases. During the first (preparatory) phase, sensitization of relevant stakeholders and recruitment of trainees will be conducted. In the second phase, formative and baseline assessment as well as training of CORNs will take place. In the third phase, which will be actual intervention phase, deployment of CORNs in their respective study site will be done and in the final phase, final evaluation and dissemination of study findings will be done. The intention behind deploying CORNs to the grassroots level is just to give a backup skilled delivery and other Maternal and Neonatal health (MNH) care services to poor rural mothers who have difficult of accessing modern health facilities for various reasons; it has no any intention to promote or encourage home deliveries or replace institutional deliveries. Perhaps it will help to assimilate rural mothers to modern health facilities. The details of the activities for each phase are discussed below.

1. Phase one : Preparatory phase At the very beginning of the intervention, sensitization and orientation workshops will be organized to be held with relevant regional and zonal level health service mangers and other concerned stakeholders on the purpose of the study. After which another workshop will also be organized with experienced and relevant experts at various capacities and responsibilities to finalize the curriculum of trainees as per the predefined core competencies of the intervention. With this developed curriculum, training manual will be prepared and recruitment of candidates sooner commences.

   Selection of candidates will be done both from the market (Unemployed nurses or midwives) and from health facilities (nurses working at health centers and hospitals , particularly from the maternal and Child Health (MCH) unit). This will be done because of the fact that during scale up of the intervention, the effect of work experience on the quality and success of the program might be an issue of concern. It should be clear that currently in Ethiopia, there is excess number of nurses trained at both government and private colleges. Selection and deployment will not cause and shortage of professionals from work place, rather it will create job opportunities for many nurses graduated but not yet employed.

   How do CORN Trainees be Selected? The selection of candidates is done by mainly by giving intake exams (both practical and theoretical) to check their favorability to complete the training followed by an oral interview to evaluate the readiness and willingness (attitude) to provide community based services at grass root level on a door to door basis. It will also help to determine the level of candidates' knowledge and clinical skills. This will be done in collaboration with Dilla University and the Southern Regional Health Bureau.
2. Phase two : Pre - Implementation Phase Having identified 16 suitable candidates (some will be in the awaiting list, not to be enrolled to the actual intervention) for the training, a four months practice oriented training will be given to them at the University's Referral Hospital and other health facilities (health centers) in the Zone.

The education of a CORN will be of good quality at both pre-service and in-service levels with a system for supportive supervision. The education of a CORN will be based on a ''Competency Model''(18). The International Confederation of Midwives (ICM) competency model is currently considered to be the international standard for provision of skilled, safe, professional care to childbearing women and their families. This model forms the conceptual framework upon which the core skills and abilities of a Skilled Birth Attendant is based reflecting essential knowledge, skills and behaviors expected during ante-partum, intra-partum, post-partum and neonatal care. Hence, the training of CORN will include critical components such as practical skills, problem solving, critical thinking and skills in decision making. These components will be thought using a large degree of student centered and facilitation approaches to teaching and learning.

After candidates have successfully completed the training acquiring the expected knowledge and skills on major core competencies; another workshop will be organized for sensitization and advocacy of the role of CORN to key influential peoples in the community (political and community leaders, mothers and other concerned bodies). In the mean time, a baseline survey will be conducted to document the coverage of skilled birth attendances and other reproductive health services across each arm of the study. Selection of clusters and study site identification will also be done during this time.

Data Collection For the baseline and end line survey (pre and post test), relevant data on: Socio-demographic characteristics, reproductive history, health seeking behavior, health service utilization, socioeconomic and socio-cultural factors affecting health service utilization ..etc will be collected using appropriate data collection tools. The tools will be pretested on 5% of study population size in non-study areas of Gedeo zone.

ETHICAL CONSIDERATION Though the proposed formative and intervention studies are non -invasive by nature, since the strategy of availing skilled birth attendants at household level is a new initiative, it may have various ethical issues.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are willing
* Permanent residents

Exclusion Criteria:

* Pregnant mother not from the selected Kebeles.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2670 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage increase in skilled Delivery | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire).
Percent of stakeholders accepting CORN intervention | 9 month
  This will be measured twice (baseline and end line qualitative survey).

SECONDARY OUTCOMES:
Percent of FP (long term)services uptake | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire).
Percent of FANC services uptake | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire).
Percent of PNC services uptake | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire).
Percent of PMTCT uptake | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire).
Neonatal morbidity | 9 month
  This will be measured twice (baseline and end line survey using interviewer administered questionnaire and from health facility records!)

CONTACTS AND LOCATIONS:
Overall Officials: Taddese Alemu, PhD, Principal Investigator — Dilla University
Locations (1):
- Dilla University, College of Medicine and Health Sciences, Addis Ababa, Ethiopia

REFERENCES:
- [Background] WHO, UNICEF, UNFPA and The World Bank, 2. Trends in maternal mortality: 1990 to 2010; Geneva, Switzerland, 2012
- [Background] Ahmed Abdella: Maternal Mortality Trend in Ethiopia, Ethiop. J. Health Dev. 2010;24 Special Issue 1:115-122
- [Background] Fauveau V, Stewart K, Khan SA, Chakraborty J. Effect on mortality of community-based maternity-care programme in rural Bangladesh. Lancet. 1991 Nov 9;338(8776):1183-6. doi: 10.1016/0140-6736(91)92041-y. PMID 1682600
- [Background] Mesganaw F, Olwit G, Shamebo D. Determinants of ANC attendance and preference to place of delivery in Gulele District. Ethiop J Health Dev. 1992;6(2):17-22
- [Background] Adegoke AA, van den Broek N. Skilled birth attendance-lessons learnt. BJOG. 2009 Oct;116(Suppl 1):33-40. doi: 10.1111/j.1471-0528.2009.02336.x. PMID 19740170
- [Background] Medhanyie A, Spigt M, Kifle Y, Schaay N, Sanders D, Blanco R, GeertJan D, Berhane Y. The role of health extension workers in improving utilization of maternal health services in rural areas in Ethiopia: a cross sectional study. BMC Health Serv Res. 2012 Oct 8;12:352. doi: 10.1186/1472-6963-12-352. PMID 23043288
- [Background] Medhanyie A, Spigt M, Dinant G, Blanco R. Knowledge and performance of the Ethiopian health extension workers on antenatal and delivery care: a cross-sectional study. Hum Resour Health. 2012 Nov 21;10:44. doi: 10.1186/1478-4491-10-44. PMID 23171076
- [Background] Mekonnen Yared, Mekonnen Asnaketch. Utilization of Maternal Health Care Services in Ethiopia. Calverton, Maryland, USA: ORC Macro; 2002
- [Background] Teferra AS, Alemu FM, Woldeyohannes SM. Institutional delivery service utilization and associated factors among mothers who gave birth in the last 12 months in Sekela District, north west of Ethiopia: a community-based cross sectional study. BMC Pregnancy Childbirth. 2012 Jul 31;12:74. doi: 10.1186/1471-2393-12-74. PMID 22849421
- [Background] Girma M, Yaya Y, Gebrehanna E, Berhane Y, Lindtjorn B. Lifesaving emergency obstetric services are inadequate in south-west Ethiopia: a formidable challenge to reducing maternal mortality in Ethiopia. BMC Health Serv Res. 2013 Nov 4;13:459. doi: 10.1186/1472-6963-13-459. PMID 24180672
- [Background] Mesfin M, Farrow J. Determinants of ANC utilization in Arsi Zone, Central Ethiopia. Ethiop J Health Dev. 1996;10(3):171-178
- [Background] Marge Koblinsky et.al: Responding to the maternal health care challenge: The Ethiopian Health Extension Program, Ethiop. Health Dev. 2010;24 Special Issue 1:105-109
- [Background] Harvey SA, Blandon YC, McCaw-Binns A, Sandino I, Urbina L, Rodriguez C, Gomez I, Ayabaca P, Djibrina S; Nicaraguan Maternal and Neonatal Health Quality Improvement Group. Are skilled birth attendants really skilled? A measurement method, some disturbing results and a potential way forward. Bull World Health Organ. 2007 Oct;85(10):783-90. doi: 10.2471/blt.06.038455. PMID 18038060
- [Background] Birhanu Z, Godesso A, Kebede Y, Gerbaba M. Mothers' experiences and satisfactions with health extension program in Jimma zone, Ethiopia: a cross sectional study. BMC Health Serv Res. 2013 Feb 21;13:74. doi: 10.1186/1472-6963-13-74. PMID 23433479
- [Background] Zhong B. How to calculate sample size in randomized controlled trial? J Thorac Dis. 2009 Dec;1(1):51-4. PMID 22263004
- [Background] MacArthur C, Winter HR, Bick DE, Knowles H, Lilford R, Henderson C, Lancashire RJ, Braunholtz DA, Gee H. Effects of redesigned community postnatal care on womens' health 4 months after birth: a cluster randomised controlled trial. Lancet. 2002 Feb 2;359(9304):378-85. doi: 10.1016/s0140-6736(02)07596-7. PMID 11844507
- [Background] Donner A, Birkett N, Buck C. Randomization by cluster. Sample size requirements and analysis. Am J Epidemiol. 1981 Dec;114(6):906-14. doi: 10.1093/oxfordjournals.aje.a113261. No abstract available. PMID 7315838
- [Background] Stanton C, Blanc AK, Croft T, Choi Y. Skilled care at birth in the developing world: progress to date and strategies for expanding coverage. J Biosoc Sci. 2007 Jan;39(1):109-20. doi: 10.1017/S0021932006001271. Epub 2006 Mar 8. PMID 16522226
- [Derived] Zerfu TA, Taddese H, Nigatu T, Tenkolu G, Khan DN, Biadgilign S, Deribew A. Is deployment of trained nurses to rural villages a remedy for the low skilled birth attendance in Ethiopia? A cluster randomized-controlled community trial. PLoS One. 2018 Oct 12;13(10):e0204986. doi: 10.1371/journal.pone.0204986. eCollection 2018. PMID 30312309
- [Derived] Zerfu TA, Ayele HT, Bogale TN. Effect of Deploying Trained Community Based Reproductive Health Nurses (CORN) on Long-Acting Reversible Contraception (LARC) Use in Rural Ethiopia: A Cluster Randomized Community Trial. Stud Fam Plann. 2018 Jun;49(2):115-126. doi: 10.1111/sifp.12054. Epub 2018 May 21. PMID 29781525
- [Derived] Zerfu TA, Taddese H, Nigatu T, Tenkolu G, Vogel JP, Khan-Neelofur D, Biadgilign S, Deribew A. Reaching the unreached through trained and skilled birth attendants in Ethiopia: a cluster randomized controlled trial study protocol. BMC Health Serv Res. 2017 Jan 26;17(1):85. doi: 10.1186/s12913-017-2041-6. PMID 28122555